CLINICAL TRIAL: NCT00025181
Title: An Open-label Study Of MDX-CTLA4 In Combination With Tyrosinase/gp100/MART-1 Peptides Emulsified With Montanide ISA 51 In The Treatment Of Patients With Resected Stage III Or Stage IV Melanoma
Brief Title: Monoclonal Antibody and Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma That Has Been Removed During Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068934 (10M-00-4); LAC-USC-10M004; MDX-MDXCTLA4-03; NCI-4210
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: iris melanoma; ciliary body and choroid melanoma, small size; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — MART-1 Antigen; incomplete Freund's adjuvant; Ipilimumab; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MART-1 antigen
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: ipilimumab
Biological: tyrosinase peptide
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Vaccines made from a person's cancer cells may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining monoclonal antibody therapy and vaccine therapy in treating patients who have stage III or stage IV melanoma that has been removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and adverse event profile of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody combined with tyrosinase:368-376, gp100:209-217, and MART-1:26-35 peptides emulsified in Montanide ISA-51 in patients with resected stage III or IV melanoma.
* Determine if this regimen causes antigen-specific T-cell activation in these patients.
* Determine the clearance profile of this regimen in these patients.
* Assess the development of host immune response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-CTLA4).

Patients receive tyrosinase:368-376, gp100:209-217, and MART-1:26-35 peptides emulsified in Montanide ISA-51 subcutaneously followed by MDX-CTLA4 IV over 90 minutes at 0, 1, 2, 3, 4, 5, 8, and 11 months in the absence of disease progression or unacceptable toxicity.

Cohorts of at least 6 patients receive escalating doses of MDX-CTLA4 until the maximum tolerated dose is determined.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter until disease progression.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed completely resected stage III or IV melanoma

  * Mucosal or ocular subtypes allowed
* HLA-A2 positive
* Positive staining of tumor tissue with antibody HMB-45 for gp100, tyrosinase, and/or MART-1
* Failed (or ineligible for or refusal of) interferon alfa

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 12 months

Hematopoietic:

* WBC at least 2,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* Hematocrit at least 30%

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 1.25 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C antibody nonreactive

Renal:

* Creatinine less than 1.25 times ULN

Immunologic:

* Antinuclear antibody (ANA) negative OR
* If ANA positive, must be:

  * Antithyroglobulin antibody negative
  * Rheumatoid factor negative
  * Anti-LKM antibody negative
  * Anti-phospholipid antibody negative
  * Anti-islet cell antibody negative
  * Anti-neutrophil cytoplasmic antibody negative
* HIV negative
* No autoimmune disease (e.g., uveitis or autoimmune inflammatory eye disease)
* No active infection
* No hypersensitivity to tyrosinase:368-376, gp100:209-217, MART-1:26-35, or Montanide ISA-51

Other:

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* No underlying medical condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody
* No prior tyrosinase, gp100, or MART-1 peptide
* No prior antitumor vaccination
* No prior interleukin-2
* At least 4 weeks since prior immunotherapy for melanoma

Chemotherapy:

* At least 4 weeks since prior chemotherapy for melanoma

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy for melanoma
* At least 4 weeks since prior corticosteroids
* No concurrent systemic or topical corticosteroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy for melanoma

Surgery:

* See Disease Characteristics

Other:

* No prior cytotoxic therapy
* At least 4 weeks since any other prior therapy for melanoma
* Concurrent analgesics allowed if on stable dose for at least 2 weeks before study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-10; Primary Completion 2003-01 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States